CLINICAL TRIAL: NCT06954597
Title: Local and Systemic Safety and Tolerability of Ascending Doses of TOP-N53, a Nitric Oxide (NO)-Releasing Phosphodiesterase-5 (PDE5) Inhibitor, Administered Topically, on Wounds in Patients With Digital Ulcers (DU) in Systemic Sclerosis (SSc) in an Open-label, Vehicle-controlled, Phase 2a, Multi-center Clinical Trial
Brief Title: Safety and Tolerability of TOP-N53 Applied on Digital Ulcers in Patients With Systemic Sclerosis
Acronym: TOP-N53-02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Topadur Pharma AG (Industry)
Collaborators: Bioskin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TOP-N53-02; 2024-511861-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-14; First posted 2025-05-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Digital Ulcers in Systemic Sclerosis
Keywords: digital ulcer; systemic sclerosis; safety; PDE5 inhibitor
MeSH Terms: conditions — digital ulcers; Scleroderma, Systemic | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: The treatment will be performed sequentially with ascending doses and treatment durations of the IMP starting with placebo treatment. The next higher dose will only be applied after safety evaluation of data of at least 2 participants per treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment step 1 (Placebo Comparator): Treatment with vehicle (= 0 µg TOP-N53), 3h exposure
  Interventions: Drug: Sildenafil; Drug: TOP-N53 vehicle
- Treatment Step 2 (Experimental): Treatment with 2 µg TOP-N53, 3h exposure
  Interventions: Drug: TOP-N53; Drug: Sildenafil
- Treatment step 3 (Experimental): Treatment with 4 µg TOP-N53, 3h exposure
  Interventions: Drug: TOP-N53; Drug: Sildenafil
- Treatment step 4 (Experimental): Treatment with 8 µg TOP-N53, 3h exposure
  Interventions: Drug: TOP-N53; Drug: Sildenafil
- Treatment step 5 (Experimental): Treatment with 8 µg TOP-N53, 24h exposure
  Interventions: Drug: TOP-N53; Drug: Sildenafil

INTERVENTIONS:
Drug: TOP-N53 — TOP-N53 solution (IMP) containing 80 µg/ml TOP-N53 is applied topically directly to the digital ulcer of patients with systemic sclerosis. The dose if defined by volume and exposure time of the IMP.
  Arms: Treatment Step 2; Treatment step 3; Treatment step 4; Treatment step 5
Drug: Sildenafil — Parallel treatment with Sildenafil 20 mg 3-times per day is permitted if patient has been on a stable dose for 2 weeks prior to screening.
Drug: TOP-N53 vehicle — TOP-N53 vehicle solution will be topically applied to digital ulcers of systemic sclerosis patients.
  Arms: Treatment step 1

SUMMARY:
The main goal of this clinical trial is to learn about how safe the new drug TOP-N53 solution is when it is applied to open wounds on the fingertip (digital ulcers) in people with an uncommon illness that results in hard, thickened areas of skin and additional problems with internal organs and blood vessels (systemic sclerosis). Another goal is to learn if different strengths of TOP-N53 can treat certain aspects of the illness. Men and women between 18 and 69 years of age with this illness may participate in the clinical trial. A parallel treatment with Sildenafil 20 mg is allowed for clinical trial participants.

The main questions the clinical trial aims to answer are:

* Does TOP-N53 cause medical problems at the fingertip wound after it is directly applied to the wound?
* Does TOP-N53 affect certain aspects of the illness like blood flow in the fingertip wounds, itch, pain, redness, bruises and bleeding at or beyond the fingertip wounds?

Researchers will compare TOP-N53 solution in different strengths to a placebo (a look-alike substance that contains no drug) to see if TOP-N53 works to affect the aspects of the illness listed above.

Participants will receive one or two treatments with the placebo or different strengths of TOP-N53. The higher strength of the drug will only be given to participants after the lower strength was found to be safe.

Participants will visit the clinic up to 8 times within a maximum of 31 days. 2 visits may be done by telephone. The doctors will ask questions to ensure that it is safe for the participants to be in the clinical trial, apply the drug and follow-up on any medical problem after the treatment. They will also test if the drug works to treat the illness by several test methods before and after the treatment. Participants will help to find out whether the drug works to treat the illness and is safe by answering questions in a diary at different timepoints before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are able to understand and follow instructions during the clinical trial.
2. Signed written informed consent in accordance with ICH-GCP and local legislation prior to admission to the clinical trial.
3. Male or female participants aged 18 to 69 years* at screening (V0) with SSc, limited or diffuse cutaneous, according to 2013 American College of Rheumatology (ACR)/EULAR criteria (*sex refers to biological characteristics).
4. At least one active DU, considered as the cardinal DU, due to SSc, ≥3 mm in diameter at screening (V0) and baseline (V1/V1b) with at least an involvement of the dermis, located at the fingertip.
5. Participants meeting one of the following 2 criteria:

   1. On stable PO sildenafil treatment at 20 mg TID [3 times per day] for at least 2 weeks prior screening (V0).
   2. Not on any PO PDE5 inhibitor (sildenafil, tadalafil, vardenafil, mirodenafil) or unselective PDE inhibitors (theophylline, dipyridamole) at any dose (including for recreational purposes) for at least 4 weeks prior screening (V0).
6. The physical examination must be without disease findings except SSc unless the investigator considers an abnormality to be irrelevant to the outcome of the clinical trial (screening [V0] and baseline [V1/V1b]).
7. Concomitant medication as endothelin receptor antagonists, calcium channel blockers, and antiplatelets must have been used at stable doses at least 2 weeks prior to screening (V0), if applicable.
8. Female volunteers of childbearing potential1 must either be permanently sterile or agree to use a highly effective birth control method (failure rate ˂1% per year when used consistently and correctly) throughout the clinical trial and for at least 7 weeks after last administration of IP.
9. A male participant with a female partner of childbearing potential1 must agree to use adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice).
10. Covered by health insurance system and/or in compliance with the recommendations of national law in force relating to biomedical research.

Exclusion Criteria:

1. Any DU accompanied by one of the following complications: Clinical infection of active ulcer/peri-ulcer, osteitis, gangrene (screening [V0] and baseline [V1/V1b]).
2. Participants with modified Rodnan Skin Score (mRSS) >35 (screening [V0]).
3. Intractable pain from DUs (NRS ≥6) (screening [V0] and baseline [V1/V1b]).
4. Active or previous history of calcinosis at the site of the designated cardinal DU.
5. Unstable organ manifestations of SSc that require immediate medical attention and treatment e.g., scleroderma renal crisis, or where other organ manifestations of SSc (interstitial lung disease [ILD], pulmonary hypertension, gastrointestinal with malabsorption syndrome or bleeding, symptomatic primary myocardial involvement) are poorly controlled and/or are determinants of clinical symptomatology.
6. Any documented active or suspected malignancy or history of malignancy within 5 years prior to the screening visit (V0), except appropriately treated basal cell carcinoma of the skin, actinic keratoses, "under surveillance" prostate cancer or in situ carcinoma of uterine cervix.
7. Participants with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment).
8. Participants with a significant disease or condition other than SSc which in the opinion of the investigator, may put the participant at risk because of participation, interfere with clinical trial procedures, or cause concern regarding the participant's ability to participate in the clinical trial or any medical condition which is expected to lead to a life expectancy <12 months.
9. Systolic BP (SBP) <95 mmHg or diastolic BP (DBP) <50 mmHg , pulse rate <50 beats per minute at sitting position (if participant is very athletic as assessed by the investigator, exception to a pulse <50 bpm is permissible) at the screening visit (V0) or baseline visit (V1/V1b); one repeat measurement will be permitted.
10. Clinically significant findings in the ECG at the screening visit (V0) or in historic ECG including 24 h Holter recordings, in particular prolongation of the QT interval corrected for HR (QTcB) ≥450 msec for men and ≥460 msec for women, ventricular arrhythmias or ectopic ventricular beats.
11. Major surgery within 8 weeks prior to the screening visit (V0).
12. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN) and total Bilirubin >1.5 x ULN.
13. Estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) formula ≤60 ml/min/1.73 m2 (corresponds to ≥ mildly to moderately reduced glomerular filtration rate [GFR]).
14. Clinical laboratory values outside the reference range that in the investigator's opinion require further investigation and preclude enrollment into the clinical trial (clinically significant).
15. Positive test for human immunodeficiency virus (HIV) antibodies, unless known from medical history.
16. Positive hepatitis B-virus surface antigen (HBsAg) test, unless known from medical history.
17. Positive anti-hepatitis C-virus antibodies (anti-HCV) test, unless known from medical history.
18. Treatment with IV prostanoids: Either ongoing, or taken in the 4 weeks before enrollment or intended for the 4 weeks after last treatment with IP during the clinical trial.
19. Treatments with PO prostanoids (selexipag), nitrovasodilators (e.g., glycerol trinitrate, isosorbide dinitrate, isosorbide mononitrate, molsidomine), soluble guanylate cyclase stimulators (riociguat) for 1 week prior screening (V0).
20. Treatment with any other PDE5 inhibitor (tadalafil, vardenafil) except sildenafil if meeting inclusion criterion no. 5a or unselective PDE inhibitor (theophylline, dipyridamole) at any posology for the 4 weeks prior screening (V0) and during the clinical trial.
21. Treatment with systemic glucocorticoids and immunosuppressants (unless used as stable background treatments for SSc at unchanged doses [as prescribed by participant's treating physicians] for at least 4 weeks prior to screening [V0]).
22. Contraindications according to the IB of sildenafil and SmPC of Sildenafil-Teva only applicable for those participants meeting inclusion criterion no 5a:

    1. Hypersensitivity to the active substance or to any of the excipients of sildenafil.
    2. Co-administration with NO donors (such as amyl nitrite) or nitrates in any form due to the hypotensive effects of nitrates.

       However, in the current clinical trial with the topical, on wound administration of the NO donor and PDE5 inhibitor TOP-N53 as IP 2 in patients on sildenafil any risk of hypotensive effects are minimal because the plasma exposure of TOP-N53 is expected as < MABEL.
    3. The co-administration of PDE5 inhibitors, including sildenafil, with guanylate cyclase stimulators, such as riociguat, is contraindicated as it may potentially lead to symptomatic hypotension.
    4. Combination with the most potent of the CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, ritonavir).
    5. Participants who have loss of vision in one eye because of non-arteritic anterior ischaemic optic neuropathy (NAION), regardless of whether this episode was in connection or not with previous PDE5 inhibitor exposure.
    6. Recent history of stroke or myocardial infarction.
23. Known or suspected hypersensitivities or known allergic reactions to components of the IPs or other dressings required for SoC during the clinical trial treatment.
24. Known allergy to local amide anesthetics.
25. Currently enrolled in another clinical investigation or clinical trial, or less than 30 days prior to screening visit (V0) (less than 2 months for any investigative clinical trials with PDE5 inhibitors, guanylate cyclase activators or stimulators, or any other intervention interfering with the broader cGMP pathway) since ending another clinical investigation or clinical trial(s), or receiving other investigational treatment(s).
26. Pregnant women or breast-feeding women.
27. In the opinion of the investigator the participant should not participate in the clinical trial if they are not expected to comply with the clinical trial protocol requirements or not expected to complete the clinical trial as scheduled.
28. Close affiliation with the investigator (e.g., a close relative) or persons working at the clinical trial center(s) or participant is an employee of sponsor(s).
29. Participant is institutionalized because of legal or regulatory order.
30. Participant is vulnerable (under legal protection).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Local treatment emergent adverse events (TEAEs) | From first treatment until Follow-up visit; up to 37 days
  Frequency of local TEAEs from treatment initiation until follow-up (FU) visit
Investigator-solicited digital ulcer (DU)-related patient reported outcome (DU-PRO) - Pain | Per dose/time escalation step at screening, at treatment days prior and several times after treatment as well as on follow-up visits during a maximum time period of 37 days.
  Frequency and mean score of pain (actual) at the cardinal DU as assessed by using a numeric rating scale (NRS, graduating intensity from 0 ['no pain'] to 10 ['worst imaginable pain']).

SECONDARY OUTCOMES:
Clinical digital ulcer (DU) assessment (CDUA) endpoint - erythema at the peri ulcer area of the cardinal DU | Per dose/time escalation step at screening, at treatment days prior and several times after treatment as well as on follow-up visits during a maximum time period of 37 days.
  Frequency and mean score of erythema at the peri ulcer area of the cardinal DU (by scoring using a 7-point Robinson scale; score 0: no reaction, score 6: worst reaction (bullous reaction or grade 3-5 reaction spreading beyounf the DU)
Clinical digital ulcer (DU) assessment (CDUA) endpoint - bruising at the peri-ulcer area of the cardinal DU or beyond | Per dose/time escalation step at screening, at treatment days prior and several times after treatment as well as on follow-up visits during a maximum time period of 37 days.
  Frequency of bruising at the peri-ulcer area of the cardinal DU or beyond (as assessed by closed question: YES/NO)
Clinical digital ulcer (DU) assessment (CDUA) endpoint - hemorrhage in the cardinal DU | Per dose/time escalation step at screening, at treatment days prior and several times after treatment as well as on follow-up visits during a maximum time period of 37 days.
  Frequency of hemorrhage in the cardinal DU (as assessed by closed question: YES/NO)
Clinical digital ulcer (DU) assessment (CDUA) endpoint - perilesional newly emerging, wound related edema at the cardinal DU | Per dose/time escalation step at screening, at treatment days prior and several times after treatment as well as on follow-up visits during a maximum time period of 37 days.
  Frequency of perilesional newly emerging, wound related edema at the cardinal DU (as assessed by closed question: YES/NO)
Clinical digital ulcer (DU) assessment (CDUA) endpoint - clinical infection at the cardinal DU | Per dose/time escalation step at screening, at treatment days prior and several times after treatment as well as on follow-up visits during a maximum time period of 37 days.
  Frequency of clinical infection at the cardinal DU (as assessed by closed question: YES/NO)
Investigator-solicited digital ulcer (DU)-related patient reported outcome (DU-PRO) - Itching | Per dose/time escalation step at screening, at treatment days prior and several times after treatment as well as on follow-up visits during a maximum time period of 37 days.
  Mean score of itching (actual) at the cardinal DU as assessed by using a numeric rating scale (NRS; graduating intensity from 0 ['no itch'] to 10 ['worst imaginable itch']).
Further investigator-solicited digital ulcer (DU) patient reported outcome (DU-PRO) | Per dose/time escalation step at 0-5 minutes after inititation of treatment and 60 minutes after removal of the IP within a time frame of up to 25 hours after IP application durng the trial period of up to 37 days.
  Number of Raynaud's phenomenon (RP) attacks since IP initiation (0-5 minutes time point) and number of RP attacks since IP removal (60 minutes time point). RP attacks are defined as episodes of reduced blood flow to the end of blood vessels usually in fingers and toes.
Systemic TEAEs | From treatment initiation until Follow-up visit; up to 37 days
  Frequency of clinically significant abnormal values for:
  * Vital signs: Mean systemic arterial blood pressure and mean pulse rate, aural body temperature (only at screening, the enrollment visit for sildenafil participants, prior IP exposure when participant arrives, and at the Follow-up visit),
  * 12 lead electrocardiogram (ECG): mean and mean changes in ECG values,
  * Safety laboratory (clinical chemistry, hematology, urinalysis, serology): mean and mean changes in laboratory values.

CONTACTS AND LOCATIONS:
Locations (5):
- France (4):
  - Centre Hospitalier Universitaire de Bordeaux, Service de Rhumatologie, Bordeaux
  - CHU Grenoble Alpes, La Tronche
  - CHRU Lille, Hôpital Claude Huriez, Rue Michel Polonosvski, Lille
  - AP-HP Hôpital Cochin, Paris
- Reha Rheinfelden, Salinenstrasse 98, Rheinfelden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No
Apart from commercially confidential information related to the IMP, data collected in the course of this clinical trial is sparse. Therefore, there is no intention to share data as no benefit for the patient community is expected by the Sponsor. This will be reconsidered if larger cohort studies are initiated in the course of the development program.